CLINICAL TRIAL: NCT01331148
Title: Pilot Study of Vitamin D to Ameliorate Chronic Pain in Sickle Cell Disease
Brief Title: High Dose Vitamin D for Sickle Cell Disease
Acronym: SCD-VitD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Children's Healthcare of Atlanta (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00014694; SCD Vitamin D (Other: Other)
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-07

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; vitamin D; pediatrics; pain
MeSH Terms: conditions — Anemia, Sickle Cell; Pain | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: randomized placebo controlled double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Active Comparator): 10,000 IU per caplet, with vitamin D dose based on weight, ranging from 240,000 IU to 600,000 IU. Patients will receive calcium/vitamin D daily soft chew as well.
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): placebo only, all patients will receive calcium/vitamin D chew
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D — 10,000 IU/caplet, patients receiving 240,000 IU to 600,000 IU cumulative Vitamin D dose based on weight.
  Other Names: cholecalciferol
  Arms: Vitamin D
Other: Placebo — placebo with daily calcium/Vitamin D soft chews
  Arms: Placebo

SUMMARY:
Vitamin D deficiency (VDD) is very common among African American adolescents and adults in the US, ten times higher than is seen in Caucasians. VDD is also quite common in sickle cell disease (SCD). Both VDD and SCD can cause chronic pain, compression fractures, and muscle weakness. The investigators believe VDD may contribute to poor musculoskeletal health and chronic pain seen in pediatric SCD. In this study, the investigators aim to show that children and adolescents with SCD and chronic pain have lower levels of vitamin D compared to those without chronic pain. The investigators also aim to determine the clinical characteristics in SCD patients related to their vitamin D status.

About 60 subjects (7 to 21 years old) will be enrolled on this study, 30 with chronic pain and 30 without chronic pain. The investigators will assess baseline characteristics including vitamin D levels, bone turnover rates (measured by C telopeptide blood levels [CTx]), markers of inflammation and oxidative stress levels in blood, baseline hemoglobin and other laboratory parameters, presence of abnormal bones on chest x-ray, pulmonary function, opioid analgesic use, overall muscle strength, quality of life and depression.

To evaluate the impact of vitamin D replacement on these baseline characteristics, the investigators will randomize subjects to receive either placebo or high dose vitamin D for 6 weeks after which time the investigators will evaluate overall vitamin D status, muscle and bone health, depression, quality of life, pain status and use of opioid pain medications, inflammation and oxidative status comparing before and after treatment with high dose vitamin D. The investigators will give-at no cost to subjects-a daily supplement that will provide the recommended daily allowance of calcium and vitamin D that contains 500mg Calcium and 200IU vitamin D to subjects throughout the study period. Subjects will be in the study for 7 months and have five to six study visits.

DETAILED DESCRIPTION:
Nearly 43% of African American adults and 53-70% of African American adolescents in the US have vitamin D deficiency (VDD), ten times more than is seen in Caucasians. VDD is also quite common in sickle cell disease (SCD) with prevalence rates of 65-100%. Pain is a hallmark symptoms of SCD accounting for the majority of SCD morbidity. Some patients with SCD develop debilitating chronic pain with an unclear etiology and unsatisfactory response to treatment. Both VDD and SCD can cause chronic pain, compression fractures and myopathy. We hypothesize that VDD is implicated in the poor musculoskeletal health and chronic pain of SCD. Therefore we aim [1] to demonstrate that pediatric sickle cell patients have high rates of VDD and those with chronic pain have lower levels of vitamin D compared to those without chronic pain [2] to evaluate the musculoskeletal health, pain status, opioid analgesic use, depression and quality of life in SCD patients with and without chronic pain and determine if the presence or severity of VDD is associated with a more severe clinical phenotype and [3] to demonstrate that administration of replacement doses of vitamin D will correct VDD, improve musculoskeletal health and ameliorate chronic pain. An additional aim of this project is to [4] evaluate and describe any correlates between vitamin D status and serum levels of inflammatory cytokines, markers of oxidative stress and vitamin D receptor polymorphisms in SCD patients with and without chronic pain.

We will evaluate 60 SCD subjects aged 7-21 years (30 with chronic pain and 30 without chronic pain) for VDD and to determine specific baseline characteristics including 25(OH)D levels, bone turnover rates measured by C telopeptide serum levels (CTx), opioid analgesic use, neuromuscular strength, evidence of skeletal complications on chest radiograph, depression and quality of life, serum levels of inflammatory cytokines and oxidative status and characteristics of the vitamin D receptor (VDR). These characteristics will be compared between those with chronic pain and those without chronic pain. We will have a 30 day run in observation period during which baseline pain status will be determined by daily pain diary report. All subjects with then be randomly assigned to receive vitamin D replacement therapy or placebo for six weeks and prospectively followed for six months. All subjects will be given daily recommended daily allowance (RDA) of calcium and vitamin D in the form of a soft chew containing 500 mg calcium and 200 IU vitamin D throughout the study period. The primary endpoints are changes in serum 25(OH)D and CTx levels and opioid analgesic use (mg/kg morphine equivalent). Secondary endpoints include changes in pain status as documented by diary, depression scores, quality of life scores, neuromuscular strength and changes in serum cytokine levels and markers of oxidative stress.

In this study we hypothesize that VDD either contributes to or exacerbates sickle cell chronic pain and that correcting VDD in SCD will result in decreased pain, depression and opioid analgesic use; an improvement in musculoskeletal health; as well as a reduction in degree of inflammation and oxidative stress. This is a pilot study in preparation for a larger prospective trial evaluating the role of VDD in the pathobiology of SCD pain and musculoskeletal health.

ELIGIBILITY:
Inclusion Criteria:

* all sickle cell genotypes including SS, SB0thal, SC, SB+Thal
* Age 7-21 years old
* Last PRBC transfusion >30 days prior

Exclusion Criteria:

* chronic renal failure
* chronic liver disease
* recent hospitalization <14 days
* history of malignancy
* serum calcium level as defined in protocol section D 2.2
* treatment with concommitant medications as defined in section D 2.2 of the protocol
* known malabsorption or short gut syndrome or conditions associated with poor GI absorption
* patients currently on high dose vitamin D therapy

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ifeyinwa Osunkwo, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12 months from study completion

REFERENCES:
- [Result] Osunkwo I, Ziegler TR, Alvarez J, McCracken C, Cherry K, Osunkwo CE, Ofori-Acquah SF, Ghosh S, Ogunbobode A, Rhodes J, Eckman JR, Dampier C, Tangpricha V. High dose vitamin D therapy for chronic pain in children and adolescents with sickle cell disease: results of a randomized double blind pilot study. Br J Haematol. 2012 Oct;159(2):211-5. doi: 10.1111/bjh.12019. Epub 2012 Aug 28. PMID 22924607

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D Arm: 10,000 IU per caplet, with vitamin D dose based on weight, ranging from 240,000 IU to 600,000 IU. Patients will receive calcium/vitamin D daily soft chew as well.
  Vitamin D: 10,000 IU/caplet, patients receiving 240,000 IU to 600,000 IU cumulative Vitamin D dose based on weight.
- Placebo Arm: placebo only, all patients will receive calcium/vitamin D chew
  Placebo: placebo with daily calcium/Vitamin D soft chews
Period: Overall Study
Arm/Group | Vitamin D Arm | Placebo Arm
Started | 23 | 23
Completed | 20 | 19
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (0.6) | 13.2 (0.8) | 13.2 (3.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 19 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 19 | 39
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
30-d pain diary pre enrollment [Mean (Standard Deviation); unit: Days with pain] — the number of days in pain during the 30 days before enrollment and start of study drug
  Days with pain | 7.7 (7.2) | 10.1 (9.7) | 8.6 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: 25 (OH)D in Nmol/L Between Baseline and 6 Months
Description: Change in 25 (OH)D level in SCD patients with and without chronic pain between baseline and 6 months.
Time Frame: Baseline and after 6 months of study participation
Population: Data for this outcome is only for completed subjects.
Measure: Mean (95% Confidence Interval); unit: nmol/L
Groups:
- Drug: Receieved Vitamin D3 supplementation and Calcium
- Placebo: Received placebo plus calcium
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 20 | 19
nmol/L | 55.2 [36.2 to 74.2] | 50.4 [29.9 to 70.9]
Statistical Analysis 1: Comparison: Drug vs Placebo; Due to the longitudinal nature of the data and presence of missing values, repeated measures analyses were conducted using the MIXED procedure in SAS. Spearman's rank correlation coefficient was used to quantify the relationship between PedsQL scores with 25OHD concentrations and pain days. Two-way analysis of variance models compared PedsQL scores between treatment groups over time; Test type: Other; p = 0.0507, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through out the 6 mo study period with a one year follow up
Description: No significant adverse events identified
Arm/Group | Vitamin D | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

LIMITATIONS AND CAVEATS:
Short follow up period small number of patients High drop out rate from adherence to diary completion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No